CLINICAL TRIAL: NCT03095274
Title: A Phase II Study of Durvalumab (MEDI4736) Plus Tremelimumab for the Treatment of Patients With Advanced Neuroendocrine Neoplasms of Gastroenteropancreatic or Lung Origin (the DUNE Trial)
Brief Title: Durvalumab (MEDI4736) Plus Tremelimumab for Advanced Neuroendocrine Neoplasms of Gastroenteropancreatic or Lung Origin
Acronym: DUNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR 15-11561-61-DUNE; 2016-002858-20 (EudraCT Number)
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Neuroendocrine Tumors; Neuroendocrine Neoplasm of Lung
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: The study includes a combined treatment of Durvalumab plus Tremelimumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Durvalumab (Experimental): Durvalumab, 1500 mg Q4W (equivalent to 20 mg/kg Q4W) for 12 months in patients ≥ 30kg.
  Weight-based dosing should be used for patients <30 kg: durvalumab 20 mg/kg.
  Interventions: Drug: Durvalumab
- Tremelimumab (Experimental): Tremelimumab 75 mg Q4W (equivalent to 1 mg/kg Q4W) for up to 4 doses/cycles in patients ≥ 30kg.
  Weight-based dosing should be used for patients <30 kg: tremelimumab 1 mg/kg Q4.
  Interventions: Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab, 1500 mg Q4W for 12 months.
  Other Names: MEDI4736
  Arms: Durvalumab
Drug: Tremelimumab — Tremelimumab 75 mg Q4W for up to 4 doses/cycles.
  Other Names: CP-675,206
  Arms: Tremelimumab

SUMMARY:
Well-differentiated gastroenteropancreatic and lung neuroendocrine tumors are generally malignancies with a prolonged natural history. However, clinical behavior is heterogeneous and when tumor progression is observed, treatment options are limited. The most used therapy for neuroendocrine tumors management are somatostatin analogs. However, even the use in lung carcinoids is quite usual, no antitumoral activity has been demonstrated. Tremelimumab and Durvalumab combination could be more efficient drugs to improve immune system activation and could obtain a significantly higher clinical benefit in these patients. Tremelimumab and Durvalumab would be the first immune combination agents showing efficacy in neuroendocrine neoplasms of different origins.

DETAILED DESCRIPTION:
Prospective, multi-center, open label, stratified, exploratory, phase II study evaluating the efficacy and safety of durvalumab plus tremelimumab in different cohorts of patients with advanced/metastatic, histologically confirmed, grade 1/2 (G1/G2) of the 2010 WHO classification neuroendocrine tumors of the pancreas, gastrointestinal tract and lung origins and grade 3 (G3) of gastroenteropancreactic system or unknown primary site (excluding lung primaries) after progression to previous therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject prior to performing any protocol-related procedures.
2. Age >18 years at time of study entry.
3. Subjects must have histologically confirmed diagnosis of one of the following advanced/metastatic neuroendocrine tumor types:

   1. Cohort 1: Well-moderately differentiated neuroendocrine tumors of the lung ( mitotic count ≤10 mitoses x 10 HPF), also known as typical and atypical lung carcinoids, that have progressed to prior somatostatin analog therapy and/or one prior targeted therapy or chemotherapy (only one prior systemic therapy, with the exception of patients that have been treated with somatostatin analogues and other systemic treatment, when two prior treatments are allowed).
   2. Cohort 2: Well-moderately differentiated G1/G2 (WHO grade 1 and 2) gastrointestinal neuroendocrine tumors after progression to somatostatin analogs and one targeted therapy (prior targeted therapy could be everolimus or a multikinase inhibitor). Prior therapies with interferon alpha-2b or radionucleotide therapy are allowed.
   3. Cohort 3: Well-moderately differentiated neuroendocrine tumors G1/G2 (WHO grade 1 and 2) from pancreatic origin after progression to standard therapies (chemotherapy, somatostatin analogs and target therapy); patients must be treated with at least two prior systemic treatment lines and a maximum of four previous treatment lines.
   4. Cohort 4: Neuroendocrine neoplasms (WHO grade 3) of gastroenteropancreatic origin of unknown primary site (excluding lung primary tumors) after progression to first-line chemotherapy with a platinum based regimen.
4. For patients included in cohorts 1, 2 and 3: WHO Classification G1/G2 (mitotic count ≤10 mitoses x 10 HPF) lung typical and atypical carcinoids for cohort 1, G1/G2 (Ki67≤20% and mitotic count ≤20 mitoses x 10 HPF) gastrointestinal for cohort 2 (including stomach, small intestine and colorectal origins), G1/G2 (Ki67≤20% and mitotic count ≤20 mitoses x 10 HPF) pancreatic for cohort 3.
5. For patients included in cohort 4: WHO classification G3 (Ki67>20% or mitotic count >20 mitoses x 10 HPF) gastroenteropancreatic neuroendocrine carcinomas (NEC) or liver metastases of G3 NEC of unknown primary site.
6. Subjects must have evidence of measurable disease meeting the following criteria:

   1. In case of more than one target lesion, it should be identified at least 1 lesion of ≥ 1.0 cm in the longest diameter for a non lymph node, or ≥ 1.5 cm in the short-axis diameter for a lymph node, which is serially measurable according to RECIST 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI). If there is only one target lesion and it is a non-lymph node, it should have a longest diameter of ≥ 1.5 cm.
   2. Lesions that have had external beam radiotherapy (EBRT) or loco-regional therapies such as radiofrequency (RF) ablation or liver embolization must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion.
   3. Subjects must show evidence of disease progression by radiologic image techniques within 12 months (an additional month will be allowed to accommodate actual dates of performance of scans, i.e., within ≤ 13 months) prior to signing informed consent, according to RECIST 1.1 .
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Life expectancy of at least 12 weeks.
9. Adequate normal organ and marrow function as defined below: Haemoglobin ≥ 9.0 g/dL; Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3); Platelet count ≥ 100 x 109/L (>100,000 per mm3).
10. Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
11. AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN.
12. Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
13. Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
14. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study.
2. Participation in another clinical study with an investigational product during the last 4 weeks.
3. WHO Classification G3 neuroendocrine neoplasms of lung origin (oat cell/large cell lung cancer).
4. Prior treatment with anti-PDL-1/anti-PD-1 or anti-CTL-4 therapy.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B (e.g., HBsAg reactive), hepatitis C (e.g., HCV RNA [qualitative] is detected) or known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
6. Known history of previous clinical diagnosis of tuberculosis.
7. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
8. Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
9. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
10. History of allogeneic organ transplant.
11. History of hypersensitivity to durvalumab, tremelimumab or any excipient.
12. Subjects having a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 28 days prior to the first dose of trial treatment.
13. Knowledge of active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they have stable brain metastases [without evidence of progression by imaging confirmed [by magnetic resonance imaging (MRI) if MRI was used at prior imaging, or confirmed by computed tomography (CT) imaging if CT used at prior imaging] for at least four weeks prior to the first dose of trial treatment; also, any neurologic symptoms must have returned to baseline], have no evidence of new or enlarging brain metastases,and have not used steroids for brain metastases for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, as subjects with carcinomatous meningitis are excluded regardless of clinical stability.
14. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab or tremelimumab. Note: The killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines, and are not allowed.
15. Subjects having known history of, or any evidence of interstitial lung disease or active, noninfectious pneumonitis.
16. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
17. Subjects who have received any anti-cancer treatment within 21 days or any investigational agent within 30 days prior to the first dose of study drug and should have recovered from any toxicity related to previous anti-cancer treatment. This does not apply to the use of somatostatin analogues for symptomatic therapy.
18. Major surgery within 3 weeks prior to the first dose of study drug.
19. Subjects having > 1+ proteinuria on urine dipstick testing will undergo 24h urine collection for quantitative assessment of proteinuria. Subjects with urine protein ≥ 1 g/24h will be ineligible.
20. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina; myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment.
21. Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction.
22. Bleeding or thrombotic disorders or use of anticoagulants, such as warfarin, or similar agents requiring therapeutic international normalized ration (INR)monitoring. Treatment with low molecular weight heparin (LMWH) is allowed.
23. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
24. Patients with tumoral disease in the head and neck region, such as paratracheal or periesophageal lymph node involvement, or with infiltration of structures in the digestive tract, or vascular pathways that represent a risk of increased bleeding.
25. Patients of cohort 1 with neuroendocrine tumors of pulmonary origin or pulmonary metastases with evidence of active bleeding.
26. Patients with evidence of digestive bleeding.
27. Active infection (any infection requiring treatment).
28. Active malignancy (except for differentiated thyroid carcinoma, or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 24 months.
29. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy or 90 days after the last dose of durvalumab monotherapy, whichever is the longer time period.
30. Documented active alcohol or drug abuse.
31. Patients with a prior history of non-compliance with medical regimens.
32. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2022-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaume Capdevila, M.D., Ph.D., Study Chair — Hospital Universitari Vall d'Hebron, Barcelona
Locations (19):
- Spain (19):
  - Instituto Catalán de Oncología Badalona, Badalona, Barcelona
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario Marqués de Valdecilla, Santander, Principality of Asturias
  - Hospital Duran i Reynals/ICO L'Hospitalet, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capdevila J, Hernando J, Teule A, Lopez C, Garcia-Carbonero R, Benavent M, Custodio A, Garcia-Alvarez A, Cubillo A, Alonso V, Carmona-Bayonas A, Alonso-Gordoa T, Crespo G, Jimenez-Fonseca P, Blanco M, Viudez A, La Casta A, Sevilla I, Segura A, Llanos M, Landolfi S, Nuciforo P, Manzano JL. Durvalumab plus tremelimumab for the treatment of advanced neuroendocrine neoplasms of gastroenteropancreatic and lung origin. Nat Commun. 2023 May 23;14(1):2973. doi: 10.1038/s41467-023-38611-5. PMID 37221181

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The DUNE study had one unique arm receiving experimental treatment (druvalumab plus tremelimumab) The DUNE trial is a multicohort study with 4 groups that have different pathologies and prognosis. Therefore, baseline characteristics and efficacy results are reported separately for each cohort.
  Please review the information in study brief summary / detailed description for further details on each cohort.
Groups:
- Durvalumab+Tremelimumab: Experiemntal: Durvalumab+Tremelimumab
  Durvalumab, 1500 mg Q4W (equivalent to 20 mg/kg Q4W) for 12 months in patients ≥ 30kg.
  Weight-based dosing should be used for patients <30 kg: durvalumab 20 mg/kg.
  Tremelimumab 75 mg Q4W (equivalent to 1 mg/kg Q4W) for up to 4 doses/cycles in patients ≥ 30kg.
  Weight-based dosing should be used for patients <30 kg: tremelimumab 1 mg/kg Q4.
Period: Overall Study
Arm/Group | Durvalumab+Tremelimumab
Started | 123
Completed | 123
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Cohort 3 : Well-moderately differentiated neuroendocrine tumors G1/G2 (WHO grade
  1 and 2) from pancreatic origin after progression to standard therapies (chemotherapy, somatostatin analogs and target therapy); patients must be treated with at least two prior systemic treatment lines and a maximum of four previous treatment lines.
Groups:
- Cohort 1 (Lung NETs): Well-moderately differentiated lung neuroendocrine tumors (classically known as typical and atypical carcinoids) after progression to somatostatin analogs and one prior targeted therapy or chemotherapy.
- Cohort 2 (G1-2 GI NENs): Well-moderately differentiated G1/G2 (WHO grade 1 and 2) gastrointestinal neuroendocrine tumors after progression to somatostatin analogs and one targeted therapy (prior targeted therapy could be everolimus or a multikinase inhibitor). Prior therapies with interferon alpha-2b or radionucleotide therapy are allowed.
- Cohort 3 (panNETs): Cohort 3 : Well-moderately differentiated neuroendocrine tumors G1/G2 (WHO grade
  1 and 2) from pancreatic origin after progression to standard therapies (chemotherapy, somatostatin analogs and target therapy); patients must be treated with at least two prior systemic treatment lines and a maximum of four previous treatment lines.
- Cohort 4 (G3 GEP NENs): Cohort 4 : Neuroendocrine neoplasms (WHO grade 3) of gastroenteropancreatic origin or unknown primary site (excluding lung primary tumors), patients will be treated in second line only, after
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Lung NETs) | Cohort 2 (G1-2 GI NENs) | Cohort 3 (panNETs) | Cohort 4 (G3 GEP NENs) | Total
Number analyzed (Participants) | 27 | 31 | 32 | 33 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.32 (11.40) | 62.77 (10.7) | 65.06 (11.29) | 56.33 (11.97) | 61.54 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 18 | 11 | 51
  Male | 18 | 18 | 14 | 22 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasic | 26 | 31 | 32 | 33 | 122
  African | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR)
Description: by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1, which is defined as the percentage of patients achieving complete response (CR), partial response (PR), or stable disease (SD) at month 9 after durvalumab plus tremelimumab was started. Assessed by Computed tomography scan (CT) or magnetic resonance imaging (MRI) CR is defined as disappearance of all target lesions; PR as >=30% decrease in the sum of the longest diameter of target lesions; SD as no changes in target lesions (i.e. <20% growth and <30% decrease). CBR = CR + PR +SD.
  Some patients were not evaluable as they had no tumor assessments.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Well-moderately differentiated lung neuroendocrine tumors (classically known as typical and atypical carcinoids) after progression to somatostatin analogs and one prior targeted therapy or chemotherapy.
- Cohort 2: Well-moderately differentiated G1/G2 (WHO grade 1 and 2) gastrointestinal neuroendocrine tumors after progression to somatostatin analogs and one targeted therapy (prior targeted therapy could be everolimus or a multikinase inhibitor). Prior therapies with interferon alpha-2b or radionucleotide therapy are allowed.
- Cohort 3: Cohort 3 : Well-moderately differentiated neuroendocrine tumors G1/G2 (WHO grade
  1 and 2) from pancreatic origin after progression to standard therapies (chemotherapy, somatostatin analogs and target therapy); patients must be treated with at least two prior systemic treatment lines and a maximum of four previous treatment lines.
- Cohort 4: Cohort 4 : Neuroendocrine neoplasms (WHO grade 3) of gastroenteropancreatic origin or unknown primary site (excluding lung primary tumors), patients will be treated in second line only, after
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 25 | 29 | 29 | 29
Participants
  CR | 0 | 0 | 0 | 1
  PR | 1 | 0 | 2 | 1
  SD | 6 | 11 | 6 | 0
  PD | 18 | 16 | 20 | 27
  Follow-up less than 9m (without previous PD/Death) | 0 | 2 | 1 | 0

2. Primary Outcome: Overall Survival
Description: Time between start of treatment and death. Here we report the median time to death from any cause, estimated by Kaplan Meier method.
  The times reported in here are the median time to event estimated by Kaplan Meier and that is why the number of months might be higher or lower than the overall and patient-specific follow-up.
Time Frame: Throughout the study period. Each patients has been followed approximately 24 months, up to 30 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 19 | 21 | 23 | 11
months | NA [NA to NA] — median not reached with the current follow.up. It is not feasible to calculate the confidence interval of a unknown (not reached) median | 29.49 [21.86 to 37.11] | 24.83 [15.33 to 34.32] | 7.04 [4.08 to 10.01]

3. Secondary Outcome: Overall Response Rate
Description: by immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) criteria.
  dAssessed by Computed tomography scan (CT) or magnetic resonance imaging (MRI) CR is defined as disappearance of all target lesions; PR as >=30% decrease in the sum of the longest diameter of target lesions. ORR = CR + PR
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 27 | 31 | 32 | 33
Participants
  CR or PR | 3 | 0 | 2 | 3
  No response | 24 | 31 | 30 | 30

4. Secondary Outcome: Duration of Response
Description: by immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) criteria.
  Assessed by Computed tomography scan (CT) or magnetic resonance imaging (MRI) CR is defined as disappearance of all target lesions; PR as >=30% decrease in the sum of the longest diameter of target lesions. Response = CR + PR
Time Frame: Throughout the study period, approximately 24 months
Population: No patient had a response to treatment (not CR, not PR)
Measure: Median (Full Range); unit: months
Groups:
- Cohort 4: Cohort 4 : Neuroendocrine neoplasms (WHO grade 3) of gastroenteropancreatic origin or unknown primary site (excluding lung primary tumors), p atients will be treated in second line only, after
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 0 | 2 | 3
months | 2.98 [2.68 to 15.50] |  | 16.31 [10.64 to 21.98] | 10.08 [3.90 to 24.26]

5. Secondary Outcome: Progression Free Survival
Description: by immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) criteria
Time Frame: Throughout the study period, approximately 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 24 | 27 | 29 | 33
months | 5.55 [4.94 to 6.17] | 5.79 [3.12 to 8.45] | 5.52 [2.38 to 8.66] | 2.41 [2.08 to 2.75]

6. Secondary Outcome: Safety - Toxicities as Defined by CTCAE, v4.0
Description: Based on subjects who experienced toxicities as defined by CTCAE, v4.0 The attribution to drug, time-of-onset, duration of the event, its resolution, and any concomitant medications.
Time Frame: 9 months
Population: In the following table, the most frequent toxicities are reported (toxicities with frequency ≥10%)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 27 | 31 | 32 | 33
Participants
  Fatigue Related: no | 19 | 16 | 12 | 21
  Fatigue Related: yes | 8 | 15 | 20 | 12
  Diarrhea Related: no | 16 | 19 | 21 | 27
  Diarrhea Related: yes | 11 | 12 | 11 | 6
  Pruritus Related: no | 23 | 21 | 22 | 28
  Pruritus Related: yes | 4 | 10 | 10 | 5
  Nausea Related: no | 26 | 25 | 24 | 30
  Nausea Related: yes | 1 | 6 | 8 | 3
  Skin and subcutaneous tissue disorders - Other, specify Related: no | 24 | 28 | 27 | 32
  Skin and subcutaneous tissue disorders - Other, specify Related: yes | 3 | 3 | 5 | 1
  Hypothyroidism Related: no | 25 | 26 | 30 | 29
  Hypothyroidism Related: yes | 2 | 5 | 2 | 4
  Vomiting Related: no | 25 | 28 | 29 | 29
  Vomiting Related: yes | 2 | 3 | 3 | 4
  Arthralgia Related: no | 25 | 27 | 26 | 32
  Arthralgia Related: yes | 2 | 4 | 6 | 1

7. Secondary Outcome: Response Status
Description: by irRECIST criteria, at 6, 9 and 12 months after start of study treatment. Assessed by Computed tomography scan (CT) or magnetic resonance imaging (MRI) CR is defined as disappearance of all target lesions; PR as >=30% decrease in the sum of the longest diameter of target lesions. ORR = CR + PR
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 27 | 31 | 32 | 33
Participants
  CR or PR | 1 | 0 | 1 | 2
  No response | 26 | 31 | 31 | 31

8. Secondary Outcome: Response Status
Description: as for outcome 7
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 27 | 31 | 32 | 33
Participants
  CR or PR | 1 | 0 | 2 | 2
  No response | 26 | 31 | 30 | 31

9. Secondary Outcome: Response Status
Description: as for outcome 7
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 27 | 31 | 32 | 33
Participants
  CR or PR | 1 | 0 | 2 | 2
  No response | 26 | 31 | 30 | 31

ADVERSE EVENTS:
Time Frame: Throughout the study period, approximately 24 months, up to 30 months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 9/27 | 17/31 | 21/32 | 30/33
Serious Adverse Events (participants affected / at risk) | 10/27 | 15/31 | 16/32 | 22/33
Other Adverse Events (participants affected / at risk) | 27/27 | 31/31 | 32/32 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=27) | Cohort 2 (N=31) | Cohort 3 (N=32) | Cohort 4 (N=33)
Abdominal pain - G2 (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain - G3 (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Acute kidney injury - G1 (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury - G3 (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury - G5 (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency - G3 (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased - G2 (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased - G3 (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anemia - G3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ascites - G5 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites - G3 (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased - G1 (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased - G3 (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Atrial fibrillation - G2 (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis - G3 (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis - G2 (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis - G3 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased - G3 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death NOS - G5 (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea - G2 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diarrhea - G3 (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Diarrhea - G4 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Diarrhea - G5 (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer - G3 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia - G3 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema limbs - G2 (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalitis infection - G5 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis G3 (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye disorders_diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue - G3 (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction G3 (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
clinical deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
GGT increased G3 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure G5 (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
trasnaminitis G2 (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cholangitis G2 (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify - G3 (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hepatitis G3 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hepatitis G4 (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis G4 (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia G3 (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia - G4 (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia - G3 (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism - G2 (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension - G2 (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism - G3 (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection G2 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction - G1 (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury to superior vena cava - G3 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis G5 (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction - G4 (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocarditis - G3 (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis - G2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis - G3 (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain - G2 (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rectal hemorrhage - G3 (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure G3 (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute renal injury G5 (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis G2 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection G3 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure - G3 (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum amylase increased - G3 (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction - G3 (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction - G5 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence - G3 (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event - G3 (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage - G3 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection - G5 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection - G2 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis G3 (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leg edemas (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visceral arterial ischemia - G5 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting - G2 (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting - G3 (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Weight loss - G1 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=27) | Cohort 2 (N=31) | Cohort 3 (N=32) | Cohort 4 (N=33)
Fatigue Grade (General disorders) | 13 (13) | 16 (16) | 20 (20) | 18 (18)
Diarrhea (Gastrointestinal disorders) | 14 (14) | 15 (15) | 12 (12) | 7 (7)
Pruritus Grade (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (11) | 11 (11) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 11 (11) | 5 (5) | 5 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 7 (7) | 3 (3) | 7 (7)
Anorexia (Metabolism and nutrition disorders) | 6 (6) | 9 (9) | 0 (0) | 7 (7)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (7) | 8 (8) | 4 (4)
Constipation Grade (Gastrointestinal disorders) | 4 (4) | 3 (3) | 9 (9) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 4 (4) | 5 (5) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (3) | 6 (6) | 3 (3)
Gastrointestinal disorders - Other, specify Grade (Gastrointestinal disorders) | 4 (4) | 7 (7) | 2 (2) | 1 (1)
Fever (General disorders) | 2 (2) | 5 (5) | 2 (2) | 5 (5)
Skin and subcutaneous tissue disorders - Other, specify Grade (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1)
Pain (Gastrointestinal disorders) | 3 (3) | 5 (5) | 4 (4) | 1 (1)
Upper respiratory infection Grade (Infections and infestations) | 4 (4) | 3 (3) | 4 (4) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 3 (3) | 6 (6) | 3 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3) | 6 (6) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 7 (7) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 3 (3) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 4 (4) | 1 (1)
Flushing Grade (Vascular disorders) | 1 (1) | 8 (8) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 3 (3) | 0 (0)
General disorders and administration site conditions (General disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Flu like symptoms (General disorders) | 2 (2) | 4 (4) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 5 (5) | 2 (2) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify Grade (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Renal and urinary disorders - Other, specify Grade (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT03095274/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03095274/SAP_001.pdf